CLINICAL TRIAL: NCT04345081
Title: Examining the Cosmetic Results and Patient Satisfaction Achieved With Skin Reducing Nipple Sparing Mastectomy of Ptotic Breast Followed by Delayed-immediate Submuscular Implant Based- Breast Reconstruction Surgery, and Comparing it to Submuscular Delayed- Immediate Implant- Based Breast Reconstruction Procedures After Skin- Sparing Mastectomy. Response-adaptive, Prospective Randomized Clinical Trial
Brief Title: Examining the Cosmetic Results, Quality of Life and Patient Satisfaction Achieved With Skin Reducing Nipple Sparing Mastectomy and Implant Based Breast Reconstruction, and Comparing it to Classic Skin- Sparing Mastectomy and Implant- Based Breast Reconstructive Surgeries
Status: Recruiting | Type: Observational
Sponsor: National Institute of Oncology, Hungary (Other)
Responsible Party: Principal Investigator, Dr. Zoltan Matrai, Head of Surgical Oncology, National Institute of Oncology, Hungary
Other Study IDs: SRNSM
Record Dates: First submitted 2020-04-05; First posted 2020-04-14 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer; Mastectomy; Lymphedema; Quality of Life; Patient Satisfaction
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SRNSM Group: Under the age of 65 with uni- or bilateral primary breast cancer ( clinical Stage 0-III), needing skin sparing mastectomy, nipple sparing mastectomy or patients require risk reducing mastectomy independently of the axillary surgery, having immediate or delayed-immediate implant based reconstruction.
  This Group receive Skin Reducing Nipple Sparing Mastectomy
  Interventions: Procedure: Skin Reducing Nipple Sparing Mastectomy and Implant Based Breast Reconstruction
- SSM Group: Under the age of 65 with uni- or bilateral primary breast cancer ( clinical Stage 0-III), needing skin sparing mastectomy, nipple sparing mastectomy or patients require risk reducing mastectomy independently of the axillary surgery, having immediate or delayed-immediate implant based reconstruction.
  This Group receive Skin Sparing Mastectomy
  Interventions: Procedure: Skin- Sparing Mastectomy and Implant- Based Breast Reconstructive Surgery

INTERVENTIONS:
Procedure: Skin Reducing Nipple Sparing Mastectomy and Implant Based Breast Reconstruction — Skin Reducing Nipple Sparing Mastectomy is performed from Inverted T incisuion and nipple is preserved.
  Groups: SRNSM Group
Procedure: Skin- Sparing Mastectomy and Implant- Based Breast Reconstructive Surgery — Classic Skin- Sparing Mastectomy
  Groups: SSM Group

SUMMARY:
This is a response-adaptive (RAR) prospective randomized study with a long-term follow-up and the aim of this clinical study is to measure with qualitative and quantitative indicators the changes in cosmetic results, quality of life and patient satisfaction after delayed- immediate breast reconstruction with standardized technique Skin Reducing Nipple sparing mastectomy, SRNSM and SSM with standardized horizontal skin incision.

According to our hypothesis, SRNSM with standardized technique on pendulous/ ptotic breasts is a safe procedure compared to SSM. It also promotes the cosmetic efficacy of SRNSM with the removal of the entire glandular tissue through avoidance of the reduction of projection, the need later nipple reconstruction surgery and of areola tattoo.

In our study we propose that compared to one of the well-known and widely investigated studied SSM, our current standardized SRNSM technique is able to perform similar oncologically safe entire gland tissue removal, with low complication rate, accommodating for adjuvant treatments. Furthermore, it may provide superior cosmetic results than SSM (NAC is not removed, projection is maintained, and there is no need for further nipple reconstruction or tattoo) with high patient satisfaction which is maintained long term.

DETAILED DESCRIPTION:
Introduction The indication of total breast removal is primarily the part of a correct oncological therapy, but secondly the removal of the full parenchyma can be prophylactic among high risk patients with positive genetic testing. In modern breast surgery, mastectomy means the removal of the entire glandular tissue. Surgery can be done in the absence of contraindication (eg. skin infiltration, mastitis carcinomatosis), by preserving the nipple-areola complex (NAC) and the skin layer above the parenchyma (nipple-sparing mastectomy, NSM) by removal of the whole or a part of the NAC (skin-sparing mastectomy, SSM) or by removal of the nipple but with the preservation of the areola (areola-sparing mastectomy, ASM). It is important to emphasize that similarly to the classic simplex mastectomy in the cases of SSM, ASM and NSM techniques provided by an experienced and qualified breast surgeon, the complete oncological removal of the mammary gland is done[1].

The essence of advanced mastectomy techniques is that they ensure the combination of radical oncological resection and immediate (immediate breast reconstruction, IBR) or delayed-immediate breast reconstructive surgery (delayed immediate breast reconstruction, D-IBR) (insertion of a tissue expander during the first operation, then as a second step replace it with a silicone implant). It avoids all the burden and negative effects of distant flap surgery, like donor scars, loss of movements etc. One or two-step post-mastectomy breast reconstructive surgeries are mainly implant-based techniques and less commonly autologous tissue techniques like distant pedicle flaps or free flaps. The tissue expander or silicone implant is placed primarily in a submuscular position but also can be inserted in a subcutaneous position in front of the large pectoral muscle. The coverage of the lower pole or even the entire surface of the implant may be strengthened with biological (so-called acellular dermal matrix) or synthetic materials (Ultrapro mesh) to reduce the pressure load of the implant on the preserved skin, the consequent skin perforation and so the loss of the implant.

The international literature of immediate or delayed-immediate postmastectomy breast reconstructive techniques is extensive and the correlation between these procedures and the oncological treatments (such as adjuvant radiotherapy) are well known [2]. According to the currently available evidence, reconstructive techniques do not adversely affect oncological outcome, so these breast surgical techniques are nowadays considered standard procedures in advanced breast cancer surgery[3]. Postmastectomy breast reconstruction surgeries are well-known as effective rehabilitation procedures, with significant psycho-oncological benefits to patients with low complication rates and high patient satisfaction. [4, 5]. Postmastectomy breast reconstructive surgery however require more sophisticated surgical techniques, special expertise, longer surgical time and significantly higher costs than simplex mastectomies.

Selecting the type of advanced mastectomy (SSM/NSM/ASM) of breast cancer depends on the location of the lesion, the size of the breast and its ptosis. Absolute contraindications of NSM are Paget disease of the nipple, bloody discharge, skin and nipple infiltration. Relative contraindications comprise pendolous/ptotic or large/larger sized breast and a distance between the nipple and tumor of less than 2cm. To achieve best cosmetic results, sparing the NAC became of prime importance, with widespread use of skin-sparing mastectomies. Sparing the skin layer and the NAC during removal of the entire glandular tissue promotes the efficiency of breast reconstruction by avoiding the reduction of projection, nipple reconstruction surgery and nipple tattoo. The cosmetic results and quality of life of those patients who had SSM instead of having NSM due to pendolous/ptotic breast are provenly unfavorable [6]. Numerous studies have proven that NSM with proper technique is an oncologically reliable method, hence it has become the part of several international protocols [7]. In the case of the high volume pendulous/ ptotic breasts, NSM and optimal implant-based breast reconstruction are achievable only by reduction of the skin-layer of the breast. The optimal surgical technique of skin-reducing nipple sparing mastectomy (SRNSM) has not been standardized yet. Due to the lack of high quality evidence and knowledge relating to the blood supply of NAC, safety of the procedure, complication rate, and oncological radicality the technique has not gained widespread popularity[8, 9].

Our present study validates the SRNSM operative technique, and also compares its results to that of classic SSM and delayed- immediate reconstruction in a response- adaptive prospective study.

Aim of the study This is a response-adaptive (RAR) [10] prospective randomized study with a long-term follow-up and the aim of this clinical study is to measure with qualitative and quantitative indicators the changes in cosmetic results, quality of life and patient satisfaction after delayed- immediate breast reconstruction with standardized technique Skin Reducing Nipple sparing mastectomy, SRNSM and SSM with standardized horizontal skin incision.

According to our hypothesis, SRNSM with standardized technique on pendulous/ ptotic breasts is a safe procedure compared to SSM. It also promotes the cosmetic efficacy of SRNSM with the removal of the entire glandular tissue through avoidance of the reduction of projection, the need later nipple reconstruction surgery and of areola tattoo.

In our study we propose that compared to one of the well-known and widely investigated studied SSM, our current standardized SRNSM technique is able to perform similar oncologically safe entire gland tissue removal, with low complication rate, accommodating for adjuvant treatments. Furthermore, it may provide superior cosmetic results than SSM (NAC is not removed, projection is maintained, and there is no need for further nipple reconstruction or tattoo) with high patient satisfaction which is maintained long term.

Patients and method Participation in the study is voluntary. In this response-adaptive (RAR) prospective randomized study, the used standardized SSM are considered to be routine procedures in the literature and in our department as well.

According to literature the SRNSM technique in not a widely used procedure. The reconstructive surgery after SSM or SRNSM do not represent new surgical procedures for our patients either in their technique nor in the indication, this prospective trial guarantee quantitative and qualitative data collection only. Applied oncological therapies are unaffected by the study and still follows the decisions of the Institute's preoperative and postoperative multidisciplinary breast cancer committee.

The study does not change the complex oncological treatment in any way compared to the institute's protocol.

Response-adaptive classification in this study means that the choice of the optimal surgical technique for the patient is not affected by the clinical trial. The selection of the surgical technique is based on the decision-making models that we use for a long time (absolute and relative contraindications), and made individually for the patient's oncological disease (eg. nipple removal), locations of the tumor, in accordance of the involvement of the skin and the existence of Paget's disease (SRNSM vs SSM), which is the same way as we treat our patients out-of-study.

Therefore, in a scientific sense, this study does not involve treatments other than routine treatment protocols.

Primary endpoint of the study:

Using correlation analysis to measure objective changes and the changes over time in oncological control, cosmetic results, quality of life and patient satisfaction achieved by different surgical techniques at one, two, three, four, and five years of follow-up.

Secondary endpoints of the study Based on the results of this study, the aim is to determine the rate of early and late postoperative complications, procedural burden (length of the operation, hospitalization).

Patients

- Under the age of 65 with uni- or bilateral primary breast cancer ( clinical Stage 0-III), needing skin sparing mastectomy, nipple sparing mastectomy or patients require risk reducing mastectomy independently of the axillary surgery, having immediate or delayed-immediate implant based reconstruction.

Exclusion criteria:

* In case the patient does not volunteer for the examination or the follow-ups
* Age above 65 years or poor general health condition, where the estimated life expectancies would be less than 2 years even without the tumorous disease
* Malignant invasive tumor in the past history (except for non-melanoma skin tumors)
* Mastectomy and reconstruction performed due pregnancy associated breast cancer
* Prior breast surgery (e.g. aesthetic surgery, mastopexy) and/or radiotherapy on the breast or in the axilla
* Malignant tumor is not removed completely with pathological examination
* Severe non-surgical (e.g. radiotherapy) complication, which could influence the aesthetic and functional results
* Autoimmune diseases
* Mastitis carcinomatosa
* Lymphangitis carcinomatosa
* Open wound therapy due SSI
* Long-term steroid usage, which changed the skin's quality and structure
* Patient under foster care, or psychically non-cooperative patient

Preoperative examination:

* Physical examination
* Triplet examination of the breast
* Chest X-ray
* Axillary ultrasound with aspiration cytology if needed
* Required additional imaging based on the oncological staging (targeted x-ray, CT, MRI, PET)
* Routine hematological and blood test analysis
* Measurements of jugulum-nipple width, nipple midline width, and nipple inframammary-fold width
* Measurement of horizontal and vertical diameter of areola
* Regnault Classification of breasts' ptosis
* Photo documentation (standard 5 directions and ap with raised arms)
* Filling out the BREAST-Q questionnaire [11]

Recorded data:

Age, weight, body mass, BMI, skin type typisation (normal, atypical, seborrheals, dehidrated, hyperhydrated (oedamatic)), preoperative cup size, presence of preoperative breast assymetry and its severity , past history, medication, smoking habits, oncological data, cTNM, pTN, pathological data, molecular genetic subtype, type of mastectomy (SM, SSM,ASM, NSM), type of primary reconstruction, neoadjuvant and adjuvant therapy, type of axillary treatment, , the size of used silicone implant(s).

Postoperative complications were classified following Clavien-Dindo Classification. [12, 13] Grade I complication does not require medication or surgical treatment (light inflammations, non-surgical haematoma or suffusion, seroma formation, partial skin/NAC loss, limited fat necrosis, SSI and lymphoedema). Grade II complication is a Grade I complication that requires medication or surgical interaction (antibiotic therapy, resuture due SSI and multiple puncture due chronic seroma). Grade III complication requires invasive surgical action (haematoma evacuation, chronic inflammation which requires reoperation, severe fat necrosis, full skin/ NAC necrosis and wound dehiscense). Grade IV complication means temporary organ failure. Grade V complication is one that leads to death.

The following data are collected in this trial: preoperative jugulum-nipple width, nipple-midline width, nipple-IMF width, vertical and horizontal width of the areola, Regnault Classification of the breast ptosis then repeating the above measurements during the follow-up (every 6 months) with parallel photo documentation and data recording of the BREAST-Q questionnaire and 5 point Likert-scale. [14]

Methods:

Enrolled patient who require unilateral SSM or SRNSM have undergone preoperative photo documentation, they filled out preoperative BREAST Q questionnaire and Regnault Classification of the breast ptosis. In case of neoadjuvant therapy, the procedure is the same and the patient selection and data recording are performed preoperatively.

The patients after modern removal of the mammary gland (SSM or SRNSM) receive adjuvant therapy based on the decision of the multidisciplinary breast cancer board of the Institute. The patients have undergone body measurements, postoperative photo documentation; they filled out postoperative BREAST Q questionnaire in the 4-6. week then 3rd and 6th months then every 6 months . Patients follow up is until the end of the 5th postoperative year.

Surgical therapy The treatment of the patients examined in the study relied on the techniques of the Breast and Sarcoma Department of the National Cancer Institute including standardized SSM in the SM control group. (See the detailed description of these: Z Mátrai, G Gulyás, T Kovács, M Kásler Principles and practice of oncoplastic breast surgery. Medicina Kiadó Zrt, 2019. 11.6. Skin-sparing and areola-sparing mastectomy) [15]

According to the valid protocol of the National Cancer Institute, the surgery of the axilla can be either sentinel lymph node biopsy or axillary lymphadenectomy/ axillary block dissection, if needed with radiotherapy of the axillary and supraclavicular region depending on the regional stage of the breast cancer. (see as well in Z Mátrai, G Gulyás, T Kovács, M Kásler Principles and practice of oncoplastic breast surgery. Medicina Kiadó Zrt, 2019. 8. fejezet: Tradicional breast surgery, 8.1.2. Axillary lymph nodee dissection; 9. Sentinel lymph node biopsy in breast cancer) [15]

See the detailed standardized techniques of immediate or delayed-immediate breast reconstruction below: Z Mátrai, G Gulyás, T Kovács, M Kásler Principles and practice of oncoplastic breast surgery. Medicina Kiadó Zrt, 2019. 11. fejezet Postmastectomy breast reconstruction, 11.4. Immediate breast reconstruction, 11.8. Subpectoral/subserratus implant based breast reconstruction) [15]

The skin reduction and the removal of the entire glandular tissue are selected according to the ptosis of the breast during SRNSM surgery.

In case of stage C-D Regnault ptosis in the upright position we mark the skin to be de-epithelialized, the footprint and the line between the midclavicular point and the nipple continuing it distally crossing the lower deflection line in accordance to stationary inverted T technique (Figure 1/A). According to the inverted T-technique, the skin reduction is carried out with gentle de-epithelization sparing the subdermal plexus. The blood supply of the nipple is secured from medial direction through the so-called medial dermal flap. Medial to the NAC, de-epithelialization should be performed with maximum sparing of subdermal plexus. (Figure 1/B) It is essential to spare the parasternal perforator vessel in the submuscular then in the subcutan space, therefore preoperative Doppler -ultrasound localization is carried out. Henceforth the removal of the entire mammary gland is performed according to the inverted T incision, with a transdermal incision from the NAC leading laterally and a supplementary T-shape incision in accordance to inverted T technique (Figure 1/C-D), standardized NSM surgery (see the detailed surgical technique below: Z Mátrai, G Gulyás, T Kovács, M Kásler Principles and practice of oncoplastic breast surgery. Medicina Kiadó Zrt, 2019. 11.7. Nipple-sparing mastectomy) [15]. It is important to note that during the removal of the entire glandular tissue and the subpectoral preparation, sparing the 2-4. perforator vessels is of high priority as these provide blood supply to the medial skin flap and thereby for the nipple. (Figure 1/E) Following the subcutaneous absorbable stitches the wound is closed by running suture. The position of the neo NAC and the preparation of the implant site on the skin layer with further de-epithelialization is determined intraoperatively; the preferable distance between the IMF and the neo nipple being 7-9 cm. (Figure 1/F)

Using and collecting cosmetic results The following data collected in standing position after marking the midline and the IMF: jugulum-nipple width, nipple-midline width and nipple-IMF width.

The breast ptosis examination performed to Regnault Classification at the beginning.

The photo documentation performed the standard way in 5 position (antero-posterior (ap), 45 degree oblique and 90 degree lateral), in ap direction both ways arms up and down with strict adherence to personal privacy policies. The patients are anonymous on the pictures without their faces, and the photo documentation performed without jewelry.

The quality of life is measured by BREAST-Q validated questionnaire. According to this, we give a score in a 1-100 scale measuring the variables of "satisfaction with the breast", "discomfort by radiotherapy", "psychosexual wellbeing" and "physical wellbeing". We use preoperatively a preoperative questionnaire and postoperatively a postoperative questionnaire. Higher rates show better quality of life [11]. The questionnaires are filled before the procedure and after the surgery in the 3rd months and every 6th months. The questionnaire is also completed by the simplex mastectomy group.

We use the Likert scale (1. definitely not, 2: no, 3: abstain, 4: agree, 4: definitely agree) for evaluating the subjective aesthetic outcome based on the photo documentation (preoperative, 4 weeks after delayed reconstruction with symmetrization, then 3rd and 6th months and every 6 months 5 years long). Based on the photo documentation three, non-involved breast surgeons make the evaluation separately without communication. The results are collected and averaged.

Follow-up:

* The follow-up is similar to the surgical and oncological follow-up in the National Cancer Institute, so it is not a burden for the patients
* The primary check-up and data registration performed preoperatively, the second check-up performed 4-6th weeks then 3rd and 6th postoperative months with photo documentation, body measurements, body mass calculation and BREAST-Q questionnaire.
* After this the photo documentation, body measurements, body mass calculation and BREAST-Q questionnaire examination performed every 6 months until the 5th year.

The bioethical background of the study:

It is a non-interventional clinical study is conducted by the competent regional research ethics committees in accordance with the Medical law 164 / A. § (2).

This non-interventional clinical trial is performed with the permission of the Ethical Committee of the National Cancer Institute according to the 23/2002. (V.9.) Medical Regulation.

The Researchers commit themselves to protect the patient's data, photo documentation in accordance with the WHO Good Clinical Practice ( based on the Helsinki Declaration) and the applicable provisions of the General Data Protection Regulation (GDPR) regarding the international ethical and scientific quality requirements pertaining to the design, conduct, documentation and reporting principles of tests conducted on humans.

Data collection and registration

- It is performed with the registration sheet for computer processing and BREAST-Q questionnaire which is an internationally validated and authorized mirror translated questionnaire. Digital photo documentation (standard 5 direction with lowered arms and ap direction with raised arms)

Planned number of patients:

The aim of the clinical study is to measure with a long-term follow-up and with qualitative and quantitative indicators the changes in cosmetic results, quality of life and patient satisfaction after delayed- immediate breast reconstruction with standardized technique Skin Reducing Nipple sparing mastectomy, SRNSM and SSM. The planned subgroups contain 50-50 cases. Planned number of patients (calculated patients' number plus 10%): 50x2=100 +10 cases

* 110 cases should be included. Planned time of patient inclusion: 1,5-2 years

Planned follow -up time:

The planned follow-up time after operation is 5 year. Interim analysis performed after 2 years median follow-up period. Final analysis is performed 5 years after closing the patient inclusion period.

ELIGIBILITY:
Inclusion Criteria:

* Under the age of 65 with uni- or bilateral primary breast cancer ( clinical Stage 0-III), needing skin sparing mastectomy, nipple sparing mastectomy or patients require risk reducing mastectomy independently of the axillary surgery, having immediate or delayed-immediate implant based reconstruction.

Exclusion Criteria:

* In case the patient does not volunteer for the examination or the follow-ups
* Age above 65 years or poor general health condition, where the estimated life expectancies would be less than 2 years even without the tumorous disease
* Malignant invasive tumor in the past history (except for non-melanoma skin tumors)
* Mastectomy and reconstruction performed due pregnancy associated breast cancer
* Prior breast surgery (e.g. aesthetic surgery, mastopexy) and/or radiotherapy on the breast or in the axilla
* Malignant tumor is not removed completely with pathological examination
* Severe non-surgical (e.g. radiotherapy) complication, which could influence the aesthetic and functional results
* Autoimmune diseases
* Mastitis carcinomatosa
* Lymphangitis carcinomatosa
* Open wound therapy due SSI
* Long-term steroid usage, which changed the skin's quality and structure
* Patient under foster care, or psychically non-cooperative patient

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The aim of the clinical study is to measure with a long-term follow-up and with qualitative and quantitative indicators the changes in cosmetic results, quality of life and patient satisfaction after delayed- immediate breast reconstruction with standardized technique Skin Reducing Nipple sparing mastectomy, SRNSM and SSM. The planned subgroups contain 50-50 cases. Planned number of patients (calculated patients' number plus 10%): 50x2=100 +10 cases
  * 110 cases should be included.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2020-04-18 (Actual); Primary Completion 2022-04-05 (Estimated); Study Completion 2027-04-05 (Estimated)

PRIMARY OUTCOMES:
Oncological safety | five years of follow-up
  Using correlation analysis to measure objective changes and the changes over time in oncological control achieved by different surgical techniques
Patients' satisfaction | five years of follow-up
  Using correlation analysis to measure objective changes and the changes over time in patients' satisfaction achieved by different surgical techniques
Cosmetic results | five years of follow-up
  Using correlation analysis to measure objective changes and the changes over time in cosmetic results achieved by different surgical techniques
Quality of life | five years of follow-up
  Using correlation analysis to measure objective changes and the changes over time in quality of life achieved by different surgical techniques

SECONDARY OUTCOMES:
Complications rate | five years of follow-up
  Based on the results of this study, the aim is to determine the rate of early and late postoperative complication.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Oncology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galimberti V, Vicini E, Corso G, Morigi C, Fontana S, Sacchini V, Veronesi P. Nipple-sparing and skin-sparing mastectomy: Review of aims, oncological safety and contraindications. Breast. 2017 Aug;34 Suppl 1(Suppl 1):S82-S84. doi: 10.1016/j.breast.2017.06.034. Epub 2017 Jun 30. PMID 28673535
- [Background] Murthy V, Chamberlain RS. Defining a place for nipple sparing mastectomy in modern breast care: an evidence based review. Breast J. 2013 Nov-Dec;19(6):571-81. doi: 10.1111/j.1524-4741.2011.01220.x. Epub 2012 Jan 29. PMID 22284266
- [Background] Weber WP, Haug M, Kurzeder C, Bjelic-Radisic V, Koller R, Reitsamer R, Fitzal F, Biazus J, Brenelli F, Urban C, Paulinelli RR, Blohmer JU, Heil J, Hoffmann J, Matrai Z, Catanuto G, Galimberti V, Gentilini O, Barry M, Hadar T, Allweis TM, Olsha O, Cardoso MJ, Gouveia PF, Rubio IT, de Boniface J, Svensjo T, Bucher S, Dubsky P, Farhadi J, Fehr MK, Fulco I, Ganz-Blattler U, Gunthert A, Harder Y, Hauser N, Kappos EA, Knauer M, Landin J, Mechera R, Meani F, Montagna G, Ritter M, Saccilotto R, Schwab FD, Steffens D, Tausch C, Zeindler J, Soysal SD, Lohsiriwat V, Kovacs T, Tansley A, Wyld L, Romics L, El-Tamer M, Pusic AL, Sacchini V, Gnant M. Oncoplastic Breast Consortium consensus conference on nipple-sparing mastectomy. Breast Cancer Res Treat. 2018 Dec;172(3):523-537. doi: 10.1007/s10549-018-4937-1. Epub 2018 Sep 4. PMID 30182349
- [Background] Rowland JH, Desmond KA, Meyerowitz BE, Belin TR, Wyatt GE, Ganz PA. Role of breast reconstructive surgery in physical and emotional outcomes among breast cancer survivors. J Natl Cancer Inst. 2000 Sep 6;92(17):1422-9. doi: 10.1093/jnci/92.17.1422. PMID 10974078
- [Background] Fang SY, Shu BC, Chang YJ. The effect of breast reconstruction surgery on body image among women after mastectomy: a meta-analysis. Breast Cancer Res Treat. 2013 Jan;137(1):13-21. doi: 10.1007/s10549-012-2349-1. Epub 2012 Dec 6. PMID 23225142
- [Background] Djohan R, Gage E, Gatherwright J, Pavri S, Firouz J, Bernard S, Yetman R. Patient satisfaction following nipple-sparing mastectomy and immediate breast reconstruction: an 8-year outcome study. Plast Reconstr Surg. 2010 Mar;125(3):818-29. doi: 10.1097/PRS.0b013e3181ccdaa4. PMID 20195110
- [Background] Morigi C. Highlights from the 15th St Gallen International Breast Cancer Conference 15-18 March, 2017, Vienna: tailored treatments for patients with early breast cancer. Ecancermedicalscience. 2017 Apr 7;11:732. doi: 10.3332/ecancer.2017.732. eCollection 2017. PMID 28491135
- [Background] Kontos M, Lanitis S, Constantinidou A, Sakarellos P, Vagios E, Tampaki EC, Tampakis A, Fragoulis M. Nipple-sparing skin-reducing mastectomy with reconstruction for large ptotic breasts. J Plast Reconstr Aesthet Surg. 2020 Apr;73(4):690-695. doi: 10.1016/j.bjps.2019.11.025. Epub 2019 Nov 28. PMID 31928958
- [Background] Falco G, Curcio A, Marongiu F, Buggi F, Mingozzi M, Mele S, Ferrari G, Folli S. Bipedicled Nipple-Sparing Mastectomy Versus Traditional Nipple-Sparing Mastectomy: Comparison of 2 Alternative Techniques in Order to Save Nipple-Areola Complex. Ann Plast Surg. 2020 Apr;84(4):366-374. doi: 10.1097/SAP.0000000000002166. PMID 31850968
- [Background] Rosenberger WF, Sverdlov O, Hu F. Adaptive randomization for clinical trials. J Biopharm Stat. 2012;22(4):719-36. doi: 10.1080/10543406.2012.676535. PMID 22651111
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Dikmans REG, Nene LEH, Bouman MB, de Vet HCW, Mureau MAM, Buncamper ME, Winters HAH, Ritt MJPF, Mullender MG. The Aesthetic Items Scale: A Tool for the Evaluation of Aesthetic Outcome after Breast Reconstruction. Plast Reconstr Surg Glob Open. 2017 Mar 1;5(3):e1254. doi: 10.1097/GOX.0000000000001254. eCollection 2017 Mar. PMID 28458968
- [Background] Mátrai Z, Gulyás G, Kovács T, et al. Principles and practice of oncoplastic breast surgery. Medicina Kiadó; 2019.